CLINICAL TRIAL: NCT00229138
Title: A Six-month, Prospective, Multicenter, Open Label, Parallel, Randomized Study of the Safety, Tolerability and Efficacy of EC-MPS With Basiliximab, Corticosteroids and Two Different Levels of Tacrolimus in de Novo Renal Transplant Recipients
Brief Title: Efficacy and Safety of Enteric-Coated Mycophenolate Sodium (EC-MPS) in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080A2409
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Kidney Transplantation
Keywords: De novo kidney recipients,; EC-MPS,; tacrolimus,; efficacy,; safety,; glomerular filtration rate; Treatment in de novo kidney recipients
MeSH Terms: interventions — Tacrolimus

ARMS (2):
- reduced Tacrolimus (Experimental)
  Interventions: Drug: EC-MPS, Tacrolimus
- Reference Tacrolimus (Active Comparator)
  Interventions: Drug: EC-MPS, Tacrolimus

INTERVENTIONS:
Drug: EC-MPS, Tacrolimus

SUMMARY:
This study will investigate the safety, tolerability and efficacy of EC-MPS with tacrolimus at both reference and reduced levels. This study will take into account safety aspects such as decreased renal toxicity by reducing the overall exposure to tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female kidney transplantation patients, 18 to 70 years of age, receiving a primary cadaveric, living unrelated, or non-HLA identical living related donor kidney.
* The renal cold ischemic time (CIT) must be <30 hours
* The age of the donor must be between 10 and 65 years

Exclusion Criteria

* Patients who have previously received an organ transplant
* Patients who are recipients of a multiple organ transplants
* Recipients of non heart-beating donor organs
* ABO incompatibility against the donor

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2005-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
renal function at 6 months posttransplant as measured by glomerular filtration rate | 6 months

SECONDARY OUTCOMES:
Efficacy as measured by combined incidence of biopsy proven acute rejection episodes, graft loss, and death at 6 months
Renal function as measured by calculated creatinine clearance
Cockcroft-Gaultand serum creatinine at 6 months
Gastrointestinal tolerability as measured by gastrointestinal
symptom rating scale (GSRS) at various time points
Safety as measured by incidence of adverse events
Effects on glucose metabolism at months 3 and 6 after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- [Result] Chan L, Andres A, Bunnapradist S, Gugliuzza K, Parasuraman R, Peddi VR, Cassuto E, Hart M. Renal Function and NODM in De Novo Renal Transplant Recipients Treated with Standard and Reduced Levels of Tacrolimus in Combination with EC-MPS. J Transplant. 2012;2012:941640. doi: 10.1155/2012/941640. Epub 2012 Nov 25. PMID 23227307